CLINICAL TRIAL: NCT05441670
Title: The Effect of a Collaborative Art Therapy and Physical Therapy Intervention on Children Undergoing a Hematopoietic Cell Transplant (HCT): a Randomized Clinical Trial
Brief Title: Art and Physical Therapy in Pediatric HCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Endowment for the Arts, United States (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 00119657; 1891731-38-22 (Other Grant/Funding Number: National Endowment of the Arts)
Record Dates: First submitted 2022-06-23; First posted 2022-07-01 (Actual); Results first posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Hematopoietic Stem Cell Transplantation; Art Therapy; Physical Therapy
MeSH Terms: interventions — Reproductive Techniques, Assisted; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Art and Physical Therapy (Experimental): 45-minutes of AT immediately followed by 30 minutes of PT Monday through Friday for 2 weeks. Targeting media that offer fluidity and tactile input, two were chosen for this study: oil pastels week 1 and gouache without brush during week 2.
  Interventions: Behavioral: Art and Physical Therapy
- Physical Therapy (Active Comparator): PT Monday through Friday for 2 weeks.
  Interventions: Behavioral: Physical Therapy

INTERVENTIONS:
Behavioral: Art and Physical Therapy — 45 minutes of Art Therapy followed by 30 minutes of Physical Therapy, Monday through Friday for 2 weeks
  Arms: Art and Physical Therapy
Behavioral: Physical Therapy — 30 minutes of Physical Therapy, Monday through Friday for 2 weeks
  Arms: Physical Therapy

SUMMARY:
The purpose of this study is to compare the effect of a combination of art therapy (AT) and physical therapy (PT) to PT only in children undergoing hematopoietic cell transplant (HCT). Each child will receive daily AT and PT or only PT for 5 days per week for 2 weeks. These sessions will begin approximately on day 15 following the transplant. Prior to starting the sessions and following 2-weeks of sessions, self-care and mobility skills will be measured. During each session, the following variables will be measured: heart rate variability (i.e., time between heart beats) using a small monitor on the chest (about the size of a quarter), walking distance using an accelerometer (similar to wearing a watch), and self-reported happiness and excitability. Although results cannot be guaranteed, it is expected that each group will benefit and demonstrate improvements in emotional state, self-care, and mobility skills.

DETAILED DESCRIPTION:
This quantitative randomized clinical trial will examine the effect of a collaborative art therapy (AT) and physical therapy (PT) intervention as compared to a PT only intervention in children undergoing a hematopoietic cell transplant. We hypothesize that physiological, emotional, selfcare, and mobility as measured by heart rate variability, Self-Assessment Manikin, walking distance and steps, and Pediatric Disability Inventory Computerized Adapted Test will demonstrate greater improvement for the AT and PT group as well as identify media that more effectively impact these physiological and health outcomes. Findings from this project may provide scientific evidence for increasing the uptake of AT and PT in children undergoing HCT.

ELIGIBILITY:
Inclusion Criteria:

* between ages 5 to 18
* Clinical Diagnosis of hematological disease
* Undergoing Hematopoietic Cell Transplantation (HCT)
* Within the inpatient hospital treatment phase of HCT

Exclusion Criteria:

* Less than age 5
* Older than age 18
* Central nervous system impairments (e.g., cerebral palsy)
* Genetic diseases (e.g., Down syndrome)
* Cognitive impairment

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Dodds, PhD, Principal Investigator — MUSC College of Health Professions
Locations (1):
- MUSC Shawn Jenkin's Children's Hospital, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scialla MA, Canter KS, Chen FF, Kolb EA, Sandler E, Wiener L, Kazak AE. Delivery of care consistent with the psychosocial standards in pediatric cancer: Current practices in the United States. Pediatr Blood Cancer. 2018 Mar;65(3):10.1002/pbc.26869. doi: 10.1002/pbc.26869. Epub 2017 Oct 28. PMID 29080381
- [Background] Jibb LA, Nathan PC, Stevens BJ, Seto E, Cafazzo JA, Stephens N, Yohannes L, Stinson JN. Psychological and Physical Interventions for the Management of Cancer-Related Pain in Pediatric and Young Adult Patients: An Integrative Review. Oncol Nurs Forum. 2015 Nov;42(6):E339-57. doi: 10.1188/15.ONF.E339-E357. PMID 26488841
- [Background] Ryan-Wenger NM. A taxonomy of children's coping strategies: a step toward theory development. Am J Orthopsychiatry. 1992 Apr;62(2):256-63. doi: 10.1037/h0079328. PMID 1580343
- [Background] Clapp LA, Taylor EP, Di Folco S, Mackinnon VL. Effectiveness of art therapy with pediatric populations affected by medical health conditions: a systematic review. Arts Health. 2019 Oct;11(3):183-201. doi: 10.1080/17533015.2018.1443952. Epub 2018 Mar 5. PMID 31038441
- [Background] Aguilar BA. The Efficacy of Art Therapy in Pediatric Oncology Patients: An Integrative Literature Review. J Pediatr Nurs. 2017 Sep-Oct;36:173-178. doi: 10.1016/j.pedn.2017.06.015. Epub 2017 Jun 30. PMID 28888499
- [Background] Newland P, Bettencourt BA. Effectiveness of mindfulness-based art therapy for symptoms of anxiety, depression, and fatigue: A systematic review and meta-analysis. Complement Ther Clin Pract. 2020 Nov;41:101246. doi: 10.1016/j.ctcp.2020.101246. Epub 2020 Oct 13. PMID 33075726
- [Background] Kuntze G, Nesbitt C, Whittaker JL, Nettel-Aguirre A, Toomey C, Esau S, Doyle-Baker PK, Shank J, Brooks J, Benseler S, Emery CA. Exercise Therapy in Juvenile Idiopathic Arthritis: A Systematic Review and Meta-Analysis. Arch Phys Med Rehabil. 2018 Jan;99(1):178-193.e1. doi: 10.1016/j.apmr.2017.05.030. Epub 2017 Jul 18. PMID 28729171
- [Background] Tang WX, Zhang LF, Ai YQ, Li ZS. Efficacy of Internet-delivered cognitive-behavioral therapy for the management of chronic pain in children and adolescents: A systematic review and meta-analysis. Medicine (Baltimore). 2018 Sep;97(36):e12061. doi: 10.1097/MD.0000000000012061. PMID 30200086
- [Background] Gonzales A, Gates E, Bhunia N, Mehyar L, Hashem H, Stanek JR, Krebs B, Auletta JJ. Transplant Energize Me Patient Outcome (TEMPO): A Quality Improvement Project that Maintains Functional Mobility in Pediatric Patients Admitted for Allogeneic Hematopoietic Cell Transplantation. Biol Blood Marrow Transplant. 2019 Sep;25(9):1779-1785. doi: 10.1016/j.bbmt.2019.05.004. Epub 2019 May 11. PMID 31085304
- [Background] Mohammed J, Smith SR, Burns L, Basak G, Aljurf M, Savani BN, Schoemans H, Peric Z, Chaudhri NA, Chigbo N, Alfred A, Bakhsh H, Salooja N, Chris Chim A, Hashmi SK. Role of Physical Therapy before and after Hematopoietic Stem Cell Transplantation: White Paper Report. Biol Blood Marrow Transplant. 2019 Jun;25(6):e191-e198. doi: 10.1016/j.bbmt.2019.01.018. Epub 2019 Jan 15. PMID 30658224
- [Background] Taverna L, Tremolada M, Bonichini S, Tosetto B, Basso G, Messina C, Pillon M. Motor skill delays in pre-school children with leukemia one year after treatment: Hematopoietic stem cell transplantation therapy as an important risk factor. PLoS One. 2017 Oct 24;12(10):e0186787. doi: 10.1371/journal.pone.0186787. eCollection 2017. PMID 29065156
- [Background] West SL, Gassas A, Schechter T, Egeler RM, Nathan PC, Wells GD. Exercise intolerance and the impact of physical activity in children treated with hematopoietic stem cell transplantation. Pediatr Exerc Sci. 2014 Aug;26(3):358-64. doi: 10.1123/pes.2013-0156. Epub 2014 Apr 10. PMID 24721685
- [Background] Carenzio G, Gherardi P, Bardoni MT, Zecca M, Bonetti F, Locatelli F, Dalla Toffola E. Rehabilitation of chronic graft versus host disease in children. A clinical series. Eura Medicophys. 2007 Dec;43(4):445-50. PMID 18084166
- [Background] Rosenhagen A, Bernhorster M, Vogt L, Weiss B, Senn A, Arndt S, Siegler K, Jung M, Bader P, Banzer W. Implementation of structured physical activity in the pediatric stem cell transplantation. Klin Padiatr. 2011 May;223(3):147-51. doi: 10.1055/s-0031-1271782. Epub 2011 Apr 1. PMID 21462101
- [Background] San Juan AF, Chamorro-Vina C, Moral S, Fernandez del Valle M, Madero L, Ramirez M, Perez M, Lucia A. Benefits of intrahospital exercise training after pediatric bone marrow transplantation. Int J Sports Med. 2008 May;29(5):439-46. doi: 10.1055/s-2007-965571. Epub 2007 Oct 25. PMID 17960520
- [Background] Chamorro-Vina C, Ruiz JR, Santana-Sosa E, Gonzalez Vicent M, Madero L, Perez M, Fleck SJ, Perez A, Ramirez M, Lucia A. Exercise during hematopoietic stem cell transplant hospitalization in children. Med Sci Sports Exerc. 2010 Jun;42(6):1045-53. doi: 10.1249/MSS.0b013e3181c4dac1. PMID 19997035
- [Background] Chamorro-Vina C, Guilcher GM, Khan FM, Mazil K, Schulte F, Wurz A, Williamson T, Reimer RA, Culos-Reed SN. EXERCISE in pediatric autologous stem cell transplant patients: a randomized controlled trial protocol. BMC Cancer. 2012 Sep 10;12:401. doi: 10.1186/1471-2407-12-401. PMID 22963378
- [Background] Rossi F, Coppo M, Zucchetti G, Bazzano D, Ricci F, Vassallo E, Nesi F, Fagioli F. Rehabilitative intervention during and after pediatric hematopoietic stem cell transplantation: An analysis of the existing literature. Pediatr Blood Cancer. 2016 Nov;63(11):1895-904. doi: 10.1002/pbc.26114. Epub 2016 Jul 13. PMID 27409063
- [Background] Jarden M, Hovgaard D, Boesen E, Quist M, Adamsen L. Pilot study of a multimodal intervention: mixed-type exercise and psychoeducation in patients undergoing allogeneic stem cell transplantation. Bone Marrow Transplant. 2007 Oct;40(8):793-800. doi: 10.1038/sj.bmt.1705807. Epub 2007 Aug 20. PMID 17704795
- [Background] Paniccia M, Paniccia D, Thomas S, Taha T, Reed N. Clinical and non-clinical depression and anxiety in young people: A scoping review on heart rate variability. Auton Neurosci. 2017 Dec;208:1-14. doi: 10.1016/j.autneu.2017.08.008. Epub 2017 Aug 26. PMID 28870754
- [Background] Kirizawa JM, Garner DM, Arab C, Valenti VE. Is heart rate variability a valuable method to investigate cardiac autonomic dysfunction in subjects with leukemia? A systematic review to evaluate its importance in clinical practice. Support Care Cancer. 2020 Jan;28(1):35-42. doi: 10.1007/s00520-019-05047-x. Epub 2019 Aug 23. PMID 31444641
- [Background] Kirizawa JM, Garner DM, Valenti VE. Impact of respiratory physical therapy on heart rate autonomic control in children with leukemia. Support Care Cancer. 2021 Mar;29(3):1585-1596. doi: 10.1007/s00520-020-05629-0. Epub 2020 Aug 1. PMID 32740892
- [Background] Porges SW. The polyvagal perspective. Biol Psychol. 2007 Feb;74(2):116-43. doi: 10.1016/j.biopsycho.2006.06.009. Epub 2006 Oct 16. PMID 17049418
- [Background] Porges SW. The polyvagal theory: new insights into adaptive reactions of the autonomic nervous system. Cleve Clin J Med. 2009 Apr;76 Suppl 2(Suppl 2):S86-90. doi: 10.3949/ccjm.76.s2.17. PMID 19376991
- [Background] Rajendra Acharya U, Paul Joseph K, Kannathal N, Lim CM, Suri JS. Heart rate variability: a review. Med Biol Eng Comput. 2006 Dec;44(12):1031-51. doi: 10.1007/s11517-006-0119-0. Epub 2006 Nov 17. PMID 17111118
- [Background] Biswas AK, Scott WA, Sommerauer JF, Luckett PM. Heart rate variability after acute traumatic brain injury in children. Crit Care Med. 2000 Dec;28(12):3907-12. doi: 10.1097/00003246-200012000-00030. PMID 11153634
- [Background] McCain GC, Ludington-Hoe SM, Swinth JY, Hadeed AJ. Heart rate variability responses of a preterm infant to kangaroo care. J Obstet Gynecol Neonatal Nurs. 2005 Nov-Dec;34(6):689-94. doi: 10.1177/0884217505281857. PMID 16282226
- [Background] Benevides TW, Lane SJ. A review of cardiac autonomic measures: considerations for examination of physiological response in children with autism spectrum disorder. J Autism Dev Disord. 2015 Feb;45(2):560-75. doi: 10.1007/s10803-013-1971-z. PMID 24154761
- [Background] Schaaf RC, Benevides TW, Leiby BE, Sendecki JA. Autonomic dysregulation during sensory stimulation in children with autism spectrum disorder. J Autism Dev Disord. 2015 Feb;45(2):461-72. doi: 10.1007/s10803-013-1924-6. PMID 23996198
- [Background] Haiblum-Itskovitch S, Czamanski-Cohen J, Galili G. Emotional Response and Changes in Heart Rate Variability Following Art-Making With Three Different Art Materials. Front Psychol. 2018 Jun 18;9:968. doi: 10.3389/fpsyg.2018.00968. eCollection 2018. PMID 29967587
- [Background] Lin YF, Lairson DR, Chan W, Du XL, Leung KS, Kennedy-Nasser AA, Martinez CA, Heslop HE, Brenner MK, Krance RA. Children with acute leukemia: a comparison of outcomes from allogeneic blood stem cell and bone marrow transplantation. Pediatr Blood Cancer. 2011 Jan;56(1):143-51. doi: 10.1002/pbc.22677. PMID 21108446
- [Background] Dumas HM, Fragala-Pinkham MA. Concurrent validity and reliability of the pediatric evaluation of disability inventory-computer adaptive test mobility domain. Pediatr Phys Ther. 2012 Summer;24(2):171-6; discussion 176. doi: 10.1097/PEP.0b013e31824c94ca. PMID 22466386
- [Background] Haley SM, Coster WJ, Dumas HM, Fragala-Pinkham MA, Kramer J, Ni P, Tian F, Kao YC, Moed R, Ludlow LH. Accuracy and precision of the Pediatric Evaluation of Disability Inventory computer-adaptive tests (PEDI-CAT). Dev Med Child Neurol. 2011 Dec;53(12):1100-6. doi: 10.1111/j.1469-8749.2011.04107.x. Epub 2011 Nov 11. PMID 22077695
- [Background] Shore BJ, Allar BG, Miller PE, Matheney TH, Snyder BD, Fragala-Pinkham M. Measuring the Reliability and Construct Validity of the Pediatric Evaluation of Disability Inventory-Computer Adaptive Test (PEDI-CAT) in Children With Cerebral Palsy. Arch Phys Med Rehabil. 2019 Jan;100(1):45-51. doi: 10.1016/j.apmr.2018.07.427. Epub 2018 Aug 18. PMID 30130519
- [Background] Fragala-Pinkham MA, Dumas HM, Lombard KA, O'Brien JE. Responsiveness of the Pediatric Evaluation of Disability Inventory-Computer Adaptive Test in measuring functional outcomes for inpatient pediatric rehabilitation. J Pediatr Rehabil Med. 2016 Sep 2;9(3):215-22. doi: 10.3233/PRM-160382. PMID 27612081
- [Background] Morinder G, Mattsson E, Sollander C, Marcus C, Larsson UE. Six-minute walk test in obese children and adolescents: reproducibility and validity. Physiother Res Int. 2009 Jun;14(2):91-104. doi: 10.1002/pri.428. PMID 19003813
- [Background] Dunaway Young S, Montes J, Kramer SS, Marra J, Salazar R, Cruz R, Chiriboga CA, Garber CE, De Vivo DC. Six-minute walk test is reliable and valid in spinal muscular atrophy. Muscle Nerve. 2016 Nov;54(5):836-842. doi: 10.1002/mus.25120. Epub 2016 May 13. PMID 27015431
- [Background] Mizrahi D, Fardell JE, Cohn RJ, Partin RE, Howell CR, Hudson MM, Robison LL, Ness KK, McBride J, Field P, Wakefield CE, Simar D. The 6-minute walk test is a good predictor of cardiorespiratory fitness in childhood cancer survivors when access to comprehensive testing is limited. Int J Cancer. 2020 Aug 1;147(3):847-855. doi: 10.1002/ijc.32819. Epub 2019 Dec 17. PMID 31800093
- [Background] Bradley MM, Lang PJ. Measuring emotion: the Self-Assessment Manikin and the Semantic Differential. J Behav Ther Exp Psychiatry. 1994 Mar;25(1):49-59. doi: 10.1016/0005-7916(94)90063-9. PMID 7962581
- [Background] McManis MH, Bradley MM, Berg WK, Cuthbert BN, Lang PJ. Emotional reactions in children: verbal, physiological, and behavioral responses to affective pictures. Psychophysiology. 2001 Mar;38(2):222-31. PMID 11347868
- [Background] Sharp C, van Goozen S, Goodyer I. Children's subjective emotional reactivity to affective pictures: gender differences and their antisocial correlates in an unselected sample of 7-11-year-olds. J Child Psychol Psychiatry. 2006 Feb;47(2):143-50. doi: 10.1111/j.1469-7610.2005.01464.x. PMID 16423145
- [Background] Murdoch M, Partin MR, Vang D, Kehle-Forbes SM. The Psychological Risk of Minimal Risk Activities: A Pre- and Posttest Study Using the Self-Assessment Manikin. J Empir Res Hum Res Ethics. 2019 Feb;14(1):15-22. doi: 10.1177/1556264618810302. Epub 2018 Nov 8. PMID 30406711
- [Background] O'Neil ME, Fragala-Pinkham MA, Forman JL, Trost SG. Measuring reliability and validity of the ActiGraph GT3X accelerometer for children with cerebral palsy: a feasibility study. J Pediatr Rehabil Med. 2014;7(3):233-40. doi: 10.3233/PRM-140292. PMID 25260506
- [Background] Hamari L, Kullberg T, Ruohonen J, Heinonen OJ, Diaz-Rodriguez N, Lilius J, Pakarinen A, Myllymaki A, Leppanen V, Salantera S. Physical activity among children: objective measurements using Fitbit One(R) and ActiGraph. BMC Res Notes. 2017 Apr 20;10(1):161. doi: 10.1186/s13104-017-2476-1. PMID 28427441
- [Background] Quintana DS, Guastella AJ, Outhred T, Hickie IB, Kemp AH. Heart rate variability is associated with emotion recognition: direct evidence for a relationship between the autonomic nervous system and social cognition. Int J Psychophysiol. 2012 Nov;86(2):168-72. doi: 10.1016/j.ijpsycho.2012.08.012. Epub 2012 Aug 30. PMID 22940643
- [Background] Ulrich S, Hildenbrand FF, Treder U, Fischler M, Keusch S, Speich R, Fasnacht M. Reference values for the 6-minute walk test in healthy children and adolescents in Switzerland. BMC Pulm Med. 2013 Aug 5;13:49. doi: 10.1186/1471-2466-13-49. PMID 23915140
- [Background] Lammers AE, Hislop AA, Flynn Y, Haworth SG. The 6-minute walk test: normal values for children of 4-11 years of age. Arch Dis Child. 2008 Jun;93(6):464-8. doi: 10.1136/adc.2007.123653. Epub 2007 Aug 3. PMID 17675356
- [Background] Li AM, Yin J, Au JT, So HK, Tsang T, Wong E, Fok TF, Ng PC. Standard reference for the six-minute-walk test in healthy children aged 7 to 16 years. Am J Respir Crit Care Med. 2007 Jul 15;176(2):174-80. doi: 10.1164/rccm.200607-883OC. Epub 2007 Apr 26. PMID 17463419

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in September of 2022. Participants were recruited from the physicians, art therapists, occupational therapists, and physical therapist, who served children undergoing hematopoietic cell transplants.
Pre-assignment Details: Participants were excluded if they were undergoing a hematopoietic cell transplant for non-malignant diagnoses.
Groups:
- AT and PT: Art and physiscal therapies provided
- PT Only: Physical therapy only provided
Period: Overall Study
Arm/Group | AT and PT | PT Only
Started | 9 | 9
Completed | 9 | 7 (Two participants completed all aspects on the intervention, but did not complete the post-test outcomes secondary to ICU admission and family social challenge.)
Not Completed | 0 | 2
Not completed — Two participants completed intervention but not post-test due to ICU admit and family challenges. | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Art and Physical Therapy | Physical Therapy | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 9 | 18
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 131.6 (56.2) | 137.7 (52.3) | 134.6 (53.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 7 | 7
  Not Hispanic or Latino | 9 | 1 | 10
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Changes in Scaled Scores of the Pediatric Evaluation of Disability Inventory - Computerized Adapted Test (PEDI-CAT)
Description: Motor function within the mobility and self-care domains of the PEDI-CAT. Scaled Scores can range from 0-100 (0=less motor function in mobility and self-care, 100=optimal motor function in mobility and self-care).
Time Frame: Pre- and post- testing before and after the 10 day intervention. Pre-testing = Day before intervention (Day 0), Post-testing = Day after intervention completion (Day 11)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Art and Physical Therapy | Physical Therapy
Number analyzed (Participants) | 9 | 9
units on a scale | 1.56 (2.35) | 2.67 (1.80)

2. Primary Outcome: Changes in Walking Distance on the 6-Minute Walk Test (6WMT)
Description: Community-based walking endurance measured by the 6-Minute Walk Test (6MWT). The 6MWT records the total distance walked in meters over 6 minutes. There is no upper limit other than physical capacity; typical values for healthy children range from approximately 400-700 meters depending on age and sex. Higher distances indicate better endurance and functional mobility, while lower distances indicate reduced endurance. This measure is widely validated in pediatric populations and predictive of cardiovascular fitness in childhood cancer survivors.
Time Frame: Pre- and post- testing before and after the 10 day intervention. Baseline day before intervention (Day 0), Day after intervention completion (Day 11)
Measure: Mean (Standard Deviation); unit: Meter
Arm/Group | Art and Physical Therapy | Physical Therapy
Number analyzed (Participants) | 9 | 9
Meter | 304.02 (122.02) | 280.87 (120.16)

3. Secondary Outcome: Changes in the Self-Assessment Manikin (SAM)
Description: A non-verbal pictorial assessment technique that directly measures the valence, arousal, and dominance associated with a person's affective reaction to a wide variety of stimuli. Each item is scored on a Likert scale ranging from 1 to 5. Valence is rated from 1(unpleasant) to 5 (pleasant) and it is expected that valence scores will increase following each intervention session. Arousal is rated from 1(calm) to 5 (excited), it is expected that arousal scores will decrease following each intervention session. Dominance is rated from 1(independent) to 5 (dependence), and it is expected that dominance scores will decrease following each intervention session.
Time Frame: Collected daily at the beginning and end of each treatment session over the 10-day intervention period. (Art and physical therapy group treatment duration = 75min, physical therapy group treatment duration = 30min)
Reporting Status: Not Posted, anticipated posting 2026-12

4. Secondary Outcome: Respiratory Sinus Arrhythmia
Time Frame: Collected daily with continuous monitoring throughout the duration of the treatment session over the 10-day intervention period. (Art and physical therapy group treatment duration = 75min, physical therapy group treatment duration = 30min)
Reporting Status: Not Posted, anticipated posting 2026-12

ADVERSE EVENTS:
Time Frame: 2 years 2 months
Arm/Group | Art and Physical Therapy | Physical Therapy
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

LIMITATIONS AND CAVEATS:
Nothing to report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-05): https://cdn.clinicaltrials.gov/large-docs/70/NCT05441670/Prot_SAP_001.pdf
  • Informed Consent Form (2024-08-07): https://cdn.clinicaltrials.gov/large-docs/70/NCT05441670/ICF_000.pdf